CLINICAL TRIAL: NCT07037784
Title: Monitoring of Physiological Parameters in Real Life in Patients Managed in Anesthesia, Rehabilitation/Intensive Care Unit and Traumatology Services, Using OXYFLEX® Biosensors Versus Standard Monitoring
Brief Title: Monitoring of Patient Physiological Parameters in Real Life Using OXYFLEX® Biosensors Versus Standard Monitoring
Acronym: OXYVIVO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-CHITS-012
Record Dates: First submitted 2025-06-06; First posted 2025-06-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Physiological Parameters
Keywords: biosensor; early warning score; real care conditions; traumatology; anesthesia; intensive care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients managed in anesthesia, rehabilitation/instensive care unit and traumatology services. (Experimental): Demonstrate the relevance of the data collected from patients treated in different hospital departments, including critical emergencies, intensive care, general intensive care units, and the operating room.
  Interventions: Other: Continuous monitoring of vital constants with OXYFLEX® biosensor.

INTERVENTIONS:
Other: Continuous monitoring of vital constants with OXYFLEX® biosensor. — The comparison of physiological data (heart rate, respiratory rate, temperature, pulse oxygen saturation, hemoglobin levels) collected by the OXYFLEX® biosensor with those obtained through standard monitoring over a maximum duration of 10 hours.

SUMMARY:
The purpose of this study is to use the OXYFLEX® device in real care conditions during the hospital management of a population of patients from various hospital services. These services include patients from the severe trauma pathway, intensive care, the polyvalent intensive care unit, and the operating room. The objective is to assess the reliability of the data collected by the OXYFLEX® biosensor compared to those obtained from standard monitoring used in these different services and conditions.

DETAILED DESCRIPTION:
The OXYFLEX® device from the Tecmoled company is a non-invasive biosensor device that allows for continuous monitoring of certain vital signs (heart rate, respiratory rate, etc.) The objectif of this research is to use this device in real care conditions during the hospital management of a patient in severe trauma care, or during anesthesia or hospitalization in the intesive care unit, by comparing the data collected by the OXYFLEX® biosensor with that obtained from standard monitoring.

Continuous multiparametric monitoring is only practiced in hospitals in intensive care units. Physiological parameters in conventional units are measured intermittently every 6 to 8 hours by the paramedical team. Studies have proven the usefulness of continuous monitoring in conventional services to reduce emergency admissions to intensive care and promote earlier intra-hospital emergency team intervention. These continuous monitoring systems, thanks to advances in technology through photoplethysmography, are becoming more affordable, miniaturized, and efficient through biosensors.

The interest in these biosensors has already been demonstrated in regular clinical practice, particularly at the Hôpital Nationale d'Instruction des Armées Sainte Anne (Guardian device), especially when coupled with alert scoring. The new OXYFLEX® biosensor, developed by the company Tecmoled, is based on a non-invasive technique of photoplethysmography, using a sensor placed on the patient's forehead with a headband. It collects pulse oxygen saturation, respiratory rate, heart rate, skin temperature, and head movements through accelerometry. It can also estimate hemoglobin concentration.

The innovative and interesting elements of this biosensor are:

* The placement on the patient's forehead, an area particularly rich in capillaries allowing for a quality signal even under pathological conditions (hypothermia, vasoconstriction).
* The number of monitored parameters, with technology continuously evolving and the future addition of new parameters (estimation of blood pressure).
* Miniaturization facilitating its use. The purpose of this research is to use this biosensor in real life to integrate it in the medium term into an early warning solution in various hospital departments (surgery department; emergency room...); and in the longer term within a project for monitoring and surveillance assisted by Artificial Intelligence in a military context, at the front.

In the current research, have been included:

* A subgroup of patients treated in the operating room for scheduled surgery, in order to test the sensors under 'ideal' conditions, that is to say, in immobile patients without failure, particularly hemodynamic.
* A subgroup of patients hospitalized in intensive care to test the sensors in more degraded conditions (hemodynamic failure, invasive mechanical ventilation...).
* A subgroup of severely traumatized patients to also test the sensor in a population of patients potentially experiencing hemodynamic failure; and requiring numerous transfers during the patient journey (emergency vital care unit,scan, angiography, operating room, intensive care...).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old);
* Patient taken care of :
* in severe traum pathway in the emergency services department
* or in the operating room for a general anesthesia procedur or locoregional anesthesia planned for a surgical duration grater than 2 hours
* or admitted to intesive care/ general intensive care units.

Exclusion Criteria:

* Opposition from the patient or their family to participate in the research ;
* Pregnant, parturient or breastfeeding woman ;
* Patient under judical protection (guardianship, curatorship …) or legal safeguarding ;
* Inability to wear the headband and the sensor (in particular : intracranial neurosurgery, othorhinolaryngology or maxillofacial surgery, debilitating trauma to the head or face …) ;
* Any other reason that, in the investigator's opinion, could interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
heart rate measurement | for a maximum of 10 hours
  The data collected by the OXYFLEX biosensor will be compared to data from standard monitoring using concordance tests, such as the Bland-Altman test, the Intraclass Correlation Coefficient (ICC), and the mean of absolute errors. These analyses will allow for the evaluation of the accuracy and reproducibility of the measurements taken with the OXYFLEX biosensor.
respiratory rate measurement | for a maximum of 10 hours
  The data collected by the OXYFLEX® biosensor will be compared to data from standard monitoring using concordance tests, such as the Bland-Altman test, the Intraclass Correlation Coefficient (ICC), and the mean of absolute errors. These analyses will allow for the evaluation of the accuracy and reproducibility of the measurements taken with the OXYFLEX® biosensor.
temperature measurement | for a maximum of 10 hours
  The data collected by the OXYFLEX® biosensor will be compared to data from standard monitoring using concordance tests, such as the Bland-Altman test, the Intraclass Correlation Coefficient (ICC), and the mean of absolute errors. These analyses will allow for the evaluation of the accuracy and reproducibility of the measurements taken with the OXYFLEX® biosensor.
pulse oxygen saturation measurement | for a maximum of 10 hours
  The data collected by the OXYFLEX® biosensor will be compared to data from standard monitoring using concordance tests, such as the Bland-Altman test, the Intraclass Correlation Coefficient (ICC), and the mean of absolute errors. These analyses will allow for the evaluation of the accuracy and reproducibility of the measurements taken with the OXYFLEX® biosensor.
hemoglobin measurement | for a maximum of 10 hours
  The data collected by the OXYFLEX® biosensor will be compared to data from standard monitoring using concordance tests, such as the Bland-Altman test, the Intraclass Correlation Coefficient (ICC), and the mean of absolute errors. These analyses will allow for the evaluation of the accuracy and reproducibility of the measurements taken with the OXYFLEX® biosensor.

SECONDARY OUTCOMES:
Conduct a clinical relevance analysis of the measurements collected by the OXYFLEX® biosensor | for a maximum of 10 hours
  The values of blood pressure will be presented as descriptive statistics (mean ± standard deviation, median, and interquartile range if necessary), but no formal statistical analysis is planned at this stage, as the objective is purely exploratory and descriptive.
Evaluate the data loss rate measured by the OXYFLEX®biosensor, based on the percentage of missing data for each parameter, in relation to the number of expected observations (per minute and/or per hour) over the total monitoring duration. | for a maximum of 10 hours
  The analysis of data loss will be based on the calculation of the percentage of missing data for each parameter, taking into account the number of observations expected to be collected per minute and the total duration of monitoring. The duration of each data loss will also be categorized (<5min, 5-14min; 15-60, 1-4 hours, >4 hours). The value of the blood pressure measured during the 10 hours of follow-up of the research will also be collected and made available for the OXYFLEX® algorithm.
Investigate the factors impacting the accuracy of measurements and the relevance of data collected by the OXYFLEX®biosensor | for a maximum of 10 hours
  Subgroup analysis of the validity of the collected data, their clinical relevance, and the technical performance of the sensor based on parameters that may alter or bias the measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- HIA Ste Anne, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No